CLINICAL TRIAL: NCT04122300
Title: Euphrasia Eye Drops in Preterm Infants With First Signs of Congestion of Nasolacrimal Duct - a Randomized Double-blind Controlled Trial
Brief Title: Euphrasia Eye Drops in Preterm Infants With First Signs of Congestion of Nasolacrimal Duct
Acronym: Euphrasia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010DR4186
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Congenita Nasolacrimal Duct Obstruction; Preterm Neonates; Ocular Discharge

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Euphrasia arm (Experimental): Euphrasia eye drops® (Weleda AG, Arlesheim) is administrated at a dose of one drop in each eye four times a day over a period of 96 hours.
  Interventions: Drug: Euphrasia Officinalis Preparation
- Placebo arm (Placebo Comparator): Placebo (0.9% NaCl) is administrated at a dose of one drop in each eye four times a day over a period of 96 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Euphrasia Officinalis Preparation — At inclusion, before the start of the therapy, a bacterial/viral and chlamydial conjunctival swab is conducted. Afterwards, both eyes of neonates are washed four times a day (i.e., every six hours) with NaCl 0.9%. Subsequently, a drop of Euphrasia is placed into the lower conjunctival sac of each eye, and followed by a lacrimal sac digital massage. If no ocular discharge is apparent for over 24 hours, the therapy is stopped. In case of worsening of symptoms or a positive swab without any improvement of symptoms an antibiotic therapy is initiated: tobramycin (Tobrex 0.3% eye drops, Novartis Pharma Switzerland). An additional swab is performed at 96 hours (i.e. at the end of the study).
  Arms: Euphrasia arm
Drug: Placebo — At inclusion, before the start of the therapy, a bacterial/viral and chlamydial conjunctival swab is conducted. Afterwards, both eyes of neonates are washed four times a day (i.e., every six hours) with NaCl 0.9%. Subsequently, a drop of placebo is placed into the lower conjunctival sac of each eye, and followed by a lacrimal sac digital massage. If no ocular discharge is apparent for over 24 hours, the therapy is stopped. In case of worsening of symptoms or a positive swab without any improvement of symptoms an antibiotic therapy is initiated: tobramycin (Tobrex 0.3% eye drops, Novartis Pharma Switzerland). An additional swab is performed at 96 hours (i.e. at the end of the study).
  Arms: Placebo arm

SUMMARY:
Congenital nasolacrimal duct obstruction (CNLDO) occurs in approximately 10 to 20% of all term newborns, and is the most common cause of persistent tearing and ocular discharge in children. CNLDO causes symptoms in up to 6% of children during the first year of life. The first clinical signs appear during the first month of life in 95% of cases and usually consist of tearing and debris on the eyelashes ("mattering"). Mucopurulent eye discharge occurs commonly in infants with CNLDO and, in the absence of other signs of infection, suggests bacterial overgrowth in the stagnant tear pool of the lacrimal sac.

This study investigates whether early administration of Euphrasia eye drops (Weleda AG, Arlesheim) in preterm neonates presenting with first ocular discharge with or without tearing and reddened eye fosters the resolution of the ocular discharge and reduces the need for topical antibiotic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates (with a gestational age of 24 to 37 weeks)
* Presenting with first signs of a congestion of the nasolacrimal duct, i.e. white, yellow, or green ocular discharge with or without tearing and reddened eye.
* Written informed consent by the parents or legal guardians

Exclusion Criteria:

* Congenital abnormalities of the eye
* Ophtalmia neonatorum
* Severe asphyxia
* Sepsis
* Intracranial bleeding (intraventricular hemorrhage ≥ grade III)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2011-05-22 (Actual); Primary Completion 2016-12-12 (Actual); Study Completion 2016-12-16 (Actual)

PRIMARY OUTCOMES:
Number of patients with treatment success at 96 hours | 96 hours
  Treatment success is defined as no ocular discharge at 96 hours and no use of topical antibiotic therapy during the 96-hour intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Wolf, Study Chair — Institute for complementary and integrative medicine
Locations (1):
- Department of Neonatology, Children University Hospital of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meier-Girard D, Gerstenberg G, Stoffel L, Kohler T, Klein SD, Eschenmoser M, Mitter VR, Nelle M, Wolf U. Euphrasia Eye Drops in Preterm Neonates With Ocular Discharge: A Randomized Double-Blind Placebo-Controlled Trial. Front Pediatr. 2020 Aug 11;8:449. doi: 10.3389/fped.2020.00449. eCollection 2020. PMID 32850558